CLINICAL TRIAL: NCT05788640
Title: Circadian and Seasonal Variation in Acute Myocardial Infarction in Relation to Blood Viscosity and Outcome Among Adults Attending the Main Assiut University Hospital
Brief Title: Circadian and Seasonal Variation in Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fady Nabil Israiel Moughiura, Resident doctor of critical care internal medicine, Assiut University
Other Study IDs: MI in seasonal variation
Record Dates: First submitted 2023-01-29; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Circadian and seasonal variation in acute myocardial infarction .

DETAILED DESCRIPTION:
Circadian and seasonal variation in acute myocardial infarction and relation between circadian rhythm and seasonal variations with biological and physiological markes of normal human being.

ELIGIBILITY:
Inclusion Criteria:

* 1.All patients above (16) years old 2.Complaint occur during acute climate changes

Exclusion Criteria:

* 1.Patients below 16 years old 2.Complaint during normal climate

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sample size was calculated using Epi- Info7. Expected frequency of cardiac onset is 15%. Based on this frequency and with a confidence limits of 6% and a confidence level of 90%, the sample needed for the study was estimated to be about from 138 patients and 196 at 95% CI .The sample will be calculated in the seasons of extreme seasonal changes at 2023, 2024
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Circadian and seasonal variation in acute myocardial infarction | Baseline
  Reporting the presence or absence of difference in electrocardiogram ,Echo and d-Dimer between patients presented with acute myocardial infarction in different seasons.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagarajan V, Fonarow GC, Ju C, Pencina M, Laskey WK, Maddox TM, Hernandez A, Bhatt DL. Seasonal and circadian variations of acute myocardial infarction: Findings from the Get With The Guidelines-Coronary Artery Disease (GWTG-CAD) program. Am Heart J. 2017 Jul;189:85-93. doi: 10.1016/j.ahj.2017.04.002. Epub 2017 Apr 12. PMID 28625385
- [Background] Thosar SS, Butler MP, Shea SA. Role of the circadian system in cardiovascular disease. J Clin Invest. 2018 Jun 1;128(6):2157-2167. doi: 10.1172/JCI80590. Epub 2018 Jun 1. PMID 29856365